CLINICAL TRIAL: NCT06227936
Title: Percutaneous Cholecystostomy, Old-fashioned or There is There Still a Role in ACC?
Brief Title: Complications of Cholecystostomy in ACC
Acronym: Chole_ACC
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: Cholecystostomy in ACC
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cholecystitis
Keywords: Acute Choleystitis; Cholecystostomy; Tokyo Guidelines; Non-Surgical Treatment; Mortality; High-risk patient
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute cholecystitis (AC) is the second most frequent pathology in Surgical Emergencies; laparoscopic cholecystectomy (LC) is the gold standard treatment, but not all patients are fit for surgery at the diagnostic. Percutaneous Cholecystostomy (PC) is an alternative to LC but has high comorbidity.

This study aims to analyse the complications of PC and review its indications in the literature.

DETAILED DESCRIPTION:
It is a single-centre retrospective study of 2000 acute cholecystitis in adults from January 2011 to december 2023, including demographyc characteristics, comorbidy severity defined as Charlson Comorbidity Index (CCI), ASA Score, Tokyo Guidelines severity classification,the indicatioons for a PC and local complications of PC.

ELIGIBILITY:
Inclusion Criteria:

* All patients admited in the Hospital del Mar with the diagnostic of an Acute Cholecystitis

Exclusion Criteria:

* Acute cholangitis
* Acute Pancreatitis
* Neoplasia
* Chronic Cholecystitis
* Patients under 18 yearls old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admited with the diagnostic of Acute Cholecystitis from January 2011 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Complications | 2011-2023
  The main outcome measure is the complications due to the PC treatment.
Mortality | 2011-2023
  The second main outcome measure is the mortality in patients with an Acute Cholecystitis and its cause.

SECONDARY OUTCOMES:
Types of cholecystostomy | 2011-2023
  There are different indications for cholecystostomy. To do a description of them.
Surgical Rescue | 2011-2023
  To study the patients that needed a surgical treatment and those who could be operated after recovery from sepsis and descrive the outcomes of all of them within the Clavien-Dindo Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González Castillo, PhD, Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No